CLINICAL TRIAL: NCT03661411
Title: Antiplatelet vs R-tPA for Acute Mild Ischemic Stroke: a Prospective, Random, Blinded Assessment of Outcome and Open Label Multi-center Study
Brief Title: Antiplatelet vs R-tPA for Acute Mild Ischemic Stroke
Acronym: ARAMIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Director, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: k（2018）22-1
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Aspirin; Clopidogrel; Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin+ clopidogrel (Experimental): aspirin 100mg qd and clopidogrel 75mg（300mg in the first day）qd with a total of 10-14 days, then oral aspirin 100mg or clopidogrel 75mg qd lasting for 90 days.
  Interventions: Drug: Aspirin; Drug: Clopidogrel 75mg
- Alteplase (Active Comparator): intravenous alteplase (0.9 mg/kg and maximal dose of 90 mg) was given, and followed by antithrombotic protocol 24 hours after thrombolysis based on clinical guideline.
  Interventions: Drug: Alteplase

INTERVENTIONS:
Drug: Aspirin — 100mg qd
  Arms: Aspirin+ clopidogrel
Drug: Clopidogrel 75mg — 75mg（after first dose of 300mg）qd
  Arms: Aspirin+ clopidogrel
Drug: Alteplase — Iv at 0.9 milligrams per kilogram (mg/kg)
  Arms: Alteplase

SUMMARY:
Acute ischemic stroke (AIS) is one of common diseases with significant morbidity, mortality and disability. A wide array of studies confirms that intravenous thrombolytic therapy with alteplase can effectively improve the functional prognosis in acute ischemic stroke. Thus all guidelines recommended the intravenous thrombolytic therapy with alteplase for acute ischemic stroke within 4.5 hours from stroke onset.

Minor stroke is usually defined as NIHSS score ≤ 3 or 5，although it accounts for 1/2-2/3 of AIS, the evidence of thrombolysis is insufficient. A study from Canada shows that 28.5% of patients with minor stroke who have not receive rt-pa thrombolytic therapy are unable to walk independently when discharged. Based on such a consideration,the PRISMS study further compares the efficacy and safety of thrombolytic therapy with antithrombotic therapy in patients with minor stroke. Unfortunately, the study has been early terminated due to the sponsorship reason in 2018, with only 313 cases enrolled. The preliminary results shows that there is no significant difference of the 90-day neurological function between the two groups, while the safety of the treatment group with alteplase has a higher rate of symptomatic intracranial hemorrhage. The patient receiving thrombolysis can not be given antithrombolytic therapy within 24 hours even if the patient's condition has worsened, is clinically more puzzling.

The CHANCE study in 2013 shows that the efficacy of aspirin with clopidogrel is superior to aspirin alone with minor stroke (NIHSS < 3) or TIA(ABCD2 < 4). The POINT study in 2018 further confirmed the efficacy and safety of intensive antithrombotic therapy within 12 hours of onset with minor stroke.

Based on the above discussion, this study aims to explore the efficacy and safety of aspirin with clopidogrel vs alteplase in the treatment of acute minor stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age ≥18 years;
2. Study treatment can be started within 4.5h;
3. Ischemic stroke confirmed by head CT or MRI;
4. NIHSS score ≤ 5, and ≤ 1 NIHSS score in single item scores such as vision, language, neglect and single limb and no score in consciousness item;
5. Premorbid mRS ≤ 1;
6. Signed informed consent

Exclusion Criteria:

1. Serious neurological deficits before onset ( mRS ≥ 2)；
2. Obvious head injuries or strokes within 3 months；
3. Subarachnoid hemorrhage;
4. History of intracranial hemorrhage;
5. Intracranial tumor, arteriovenous malformation or aneurysm;
6. Intracranial or spinal cord surgery within 3 months;
7. Arterial puncture at a noncompressible site within the previous seven days;
8. Gastrointestinal or urinary tract hemorrhage within the previous 21 days;
9. Major surgery within 1 month;
10. Systolic pressure ≥180 mmHg or diastolic pressure ≥110 mmHg;
11. Blood glucose < 50 mg/dl (2.7mmol/L);
12. Heparin therapy or oral anticoagulation therapy within 48 hours;
13. Platelet count of <100,000/mm3 (This does not need to be verified prior to randomization if clinical abnormality is not suspected);
14. Oral warfarin is being taken and INR>1.6;
15. Abnormal APTT;
16. Pregnancy;
17. Neurological deficit after epileptic seizures;
18. Myocardial infarction within 3 months;
19. Cerebral infarction with definite anticoagulation indications, such as cerebral infarction caused by cardiogenic embolism;
20. Oral administration is not allowed due to dysphagia;
21. allergy to study drugs;
22. Other serious illness that would confound the clinical outcome at 90 days;
23. Participating in other clinical trials within 3 months;
24. patients not suitable for this clinical studies considered by researcher;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 760 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-07-18 (Actual)

PRIMARY OUTCOMES:
Proportion of mRS (0-1） | 90±7 days

SECONDARY OUTCOMES:
Proportion of mRS (0-2） | 90±7 days
change in NIH Stroke Scale score compared with baseline | 24 hours
incidence of early neurological improvement | 24 hours
  more than 2 NIH Stroke Scale score decrease compared with baseline
Incidence of early neurological deterioration | 7 days
  more than 2 NIH Stroke Scale score increase (not result of cerebral hemorrhage) compared with baseline
occurrence of stroke or other vascular events | 90±7 days
proportion of death of any cause | 90±7 days
occurrence of symptomatic intracranial hemorrhage | 90±7 days
  more than 4 NIHSS score increase caused by intracranial hemorrhage
proportion of any bleeding events | 90±7 days

CONTACTS AND LOCATIONS:
Overall Officials: Huisheng Chen, Doctor, Study Chair — Neurology Department
Locations (1):
- Lin Tao, Shenyang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yao ZG, Pei YF, Chen HS. Onset to Treatment Time and Early Neurological Deterioration of Dual Antiplatelet Therapy Versus Alteplase in Minor Stroke. J Am Heart Assoc. 2025 Nov 4;14(21):e043980. doi: 10.1161/JAHA.125.043980. Epub 2025 Oct 23. PMID 41128284
- [Derived] Fei ZX, Yin Y, Cui Y, Nguyen TN, Chen HS. Dual Antiplatelet Therapy Versus Alteplase for Mild Stroke with Admission NIHSS Score 0-3 Versus 4-5: A Secondary Analysis of the ARAMIS Randomized Trial. CNS Drugs. 2025 Oct;39(10):1037-1046. doi: 10.1007/s40263-025-01211-6. Epub 2025 Aug 4. PMID 40760234
- [Derived] He XY, He C, Chen HS. Renal function and efficacy of dual antiplatelet vs. alteplase in minor stroke: a post hoc analysis of ARAMIS study. Front Neurol. 2025 Apr 30;16:1568711. doi: 10.3389/fneur.2025.1568711. eCollection 2025. PMID 40371069
- [Derived] Cui Y, Chen HS. Dual antiplatelet versus alteplase in anterior and posterior circulation minor stroke. Stroke Vasc Neurol. 2025 Aug 26;10(4):491-498. doi: 10.1136/svn-2024-003705. PMID 39663175
- [Derived] Cui Y, He C, Li ZA, Wang Y, Chen HS. Dual Antiplatelet Versus Alteplase for Early Neurologic Deterioration in Minor Stroke With Versus Without Large Vessel Occlusion: Prespecified Post Hoc Analysis of the ARAMIS Trial. Stroke. 2024 Nov;55(11):2590-2598. doi: 10.1161/STROKEAHA.124.048248. Epub 2024 Oct 10. PMID 39387110
- [Derived] Cui Y, Zhao ZA, Wang JQ, Qiu SQ, Shen XY, Li ZY, Hu HZ, Chen HS. Systolic blood pressure and early neurological deterioration in minor stroke: A post hoc analysis of ARAMIS trial. CNS Neurosci Ther. 2024 Jul;30(7):e14868. doi: 10.1111/cns.14868. PMID 39014552
- [Derived] Chen HS, Cui Y, Zhou ZH, Zhang H, Wang LX, Wang WZ, Shen LY, Guo LY, Wang EQ, Wang RX, Han J, Dong YL, Li J, Lin YZ, Yang QC, Zhang L, Li JY, Wang J, Xia L, Ma GB, Lu J, Jiang CH, Huang SM, Wan LS, Piao XY, Li Z, Li YS, Yang KH, Wang DL, Nguyen TN; ARAMIS Investigators. Dual Antiplatelet Therapy vs Alteplase for Patients With Minor Nondisabling Acute Ischemic Stroke: The ARAMIS Randomized Clinical Trial. JAMA. 2023 Jun 27;329(24):2135-2144. doi: 10.1001/jama.2023.7827. PMID 37367978